CLINICAL TRIAL: NCT07369817
Title: Optimization and Testing of ALRITE, a Clinical Decision Support Tool for Management of Respiratory Illnesses in Young Children in Primary Care Health Facilities in Uganda
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Laura Ellington, Assistant Professor, Department of Pediatrics, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00020447; 5K23HL163321-02 (NIH)
Record Dates: First submitted 2026-01-21; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Pneumonia Childhood; Childhood Asthma; Acute Lower Respiratory Illness; Wheezing Lower Respiratory Illness

STUDY DESIGN:
Intervention Model Description: Interrupted time series design, no comparison group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ALRITE deployment (Experimental): Healthcare workers will undergo training in the mobile health decision support tool called ALRITE. They will each receive an ALRITE-enabled tablet to use in clinical care. ALRITE use is encouraged but not required. Researchers will collect clinical data from the health record at each study site to evaluate the effect of the ALRITE intervention on acute lower respiratory illness diagnosis and treatment.
  Interventions: Other: ALRITE

INTERVENTIONS:
Other: ALRITE — ALRITE is a point-of-care mobile health clinical decision support tool designed for use by healthcare workers in Uganda. ALRITE guides the user into entering patient information and provides guideline-concordant recommendations. ALRITE also includes educational videos and weight-based dosing.

SUMMARY:
The goal of this study is to pilot test the feasibility of a mobile health clinical decision support tool called ALRITE for the diagnosis and management of acute lower respiratory illnesses in young children in Uganda. Asthma/wheezing illness, in particular, is underdiagnosed in this setting. The main questions the study aims to answer are:

* Are the intervention structure, processes, outcomes, and implementations strategies feasible to conduct in the desired settings?
* Does ALRITE increase the diagnosis of wheezing illness among children seen at Ugandan health centers?

Researchers will compare outcomes before and after ALRITE deployment to healthcare workers at 4 Ugandan healthcare centers using an interrupted time series design. Study participants are healthcare workers.

There will be12 months of baseline data collection ("baseline period"), at the beginning of which healthcare workers will be enrolled at each site. Following the baseline period, health workers will receive ALRITE training and will be encouraged but not required to use ALRITE in clinical care for a 6-month intervention period. Health worker participants will fill out surveys and participate in focus group discussions to provide feedback.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare workers employed at each study site with a minimum of 6 months' experience of caring for children with respiratory symptoms in general outpatient care
* Completed one of the following training programs: medical officer, clinical officer, nurse, midwife
* proficient in reading and speaking English, one of the official languages of Uganda
* at least 18 years of age

Exclusion Criteria:

* inability to read/write English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Healthcare worker enrollment (study feasibility) | At enrollment
  Number of healthcare workers enrolled during the baseline phase and additional healthcare workers who were enrolled during the remaining study period (ex: new hires or transfers)
Healthcare worker retention (study feasibility) | From enrollment through study completion, an average of 20 months
  Proportion of healthcare workers active in the study over total number enrolled
Availability of ALRITE-enabled devices (study feasibility) | Monthly during the intervention period from ALRITE deployment through study completion, an average of 6 months
  Proportion of functional devices over number of devices provided to the facility per month
ALRITE training completion (study feasibility) | During ALRITE deployment at the end of the baseline period, estimated 1-2 months
  Number of ALRITE training sessions completed per site
Data completeness (study feasibility) | Monthly from baseline (day 1) through the study completion, estimated 20 months
  Percentage of eligible pediatric cases correctly abstracted from the health facility records into the electronic database.

SECONDARY OUTCOMES:
Diagnosis rate of wheezing illness | Monthly from baseline through study completion, estimated 20 months
  Diagnosis rates of wheezing illness/asthma among all young children presenting to study sites, as recorded in the health record
Diagnosis rate of pneumonia | Monthly from baseline through study completion, estimated 20 months
  Diagnosis rates of pneumonia among all young children presenting to study sites, as recorded in the health record

CONTACTS AND LOCATIONS:
Overall Officials: Laura Ellington, MD, MS, Principal Investigator — University of Washington
Locations (1):
- Makerere University Lung Institute, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No